CLINICAL TRIAL: NCT00000200
Title: Cocaine Effects in Humans: Physiology and Behavior
Brief Title: Cocaine Effects in Humans: Physiology and Behavior - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-03818-1; R01-03818-1
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-10

CONDITIONS: Cocaine-Related Disorders
Keywords: self-administration
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Methadone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Methadone — normal maintenance dose

SUMMARY:
The purpose of this study is to compare the effects of buprenorphine or methadone maintenance on cocaine taking and on the physiological and subjective effects of cocaine, including cocaine craving, in opiate-dependent cocaine users.

ELIGIBILITY:
Please contact site for information.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 1997-01; Primary Completion 1998-01 (Actual); Study Completion 1998-01 (Actual)

PRIMARY OUTCOMES:
Interaction of cocaine and meds on cardio | 3 hr
Interaction of cocaine & meds on coc's subjective | 3 hr
Effects of medication on cocaine craving | 3 hr

CONTACTS AND LOCATIONS:
Overall Officials: Marian Fischman, Ph.D., Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

REFERENCES:
- [Result] Foltin RW, Fischman MW. Effects of methadone or buprenorphine maintenance on the subjective and reinforcing effects of intravenous cocaine in humans. J Pharmacol Exp Ther. 1996 Sep;278(3):1153-64. PMID 8819498